CLINICAL TRIAL: NCT03137589
Title: Telemedical, Intersectoral Network as New Digital Health Structure to Measurably Improve the Local Health Care
Acronym: TELnet@NRW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-162
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-01

CONDITIONS: Infection; Intensive Care Patients
Keywords: Telemedicine
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Stepped-Wedge-Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients of this group are routinely treated without telemedical support.
- Telemedical support (Active Comparator): Patients of this group are routinely treated with telemedical support.
  Interventions: Other: Telemedical support

INTERVENTIONS:
Other: Telemedical support — Participating sites will be advised by telemedicine support.
  Arms: Telemedical support

SUMMARY:
Telemedicine allows providing expert know-ledge from specialized health centers to regional hospitals and practices. In this multicenter, prospective, non-interventional study hospitals and practices in NRW are supplied via a telematics platform with expertise from the university hospitals RWTH Aachen and Münster. The communication occurs via highly encrypted audio/video conference systems and a certified data exchange platform "Fallakte+". In total 40.000 outpatient and stationary patients with infectious diseases or need for intensive care should be treated with telemedical support. The participating hospitals and practices are randomly distributed into four clusters. The clusters are supplied with telemedicine at different time points but all clusters start at the same time collecting data from patient cohorts of infectiology and intensive care (e.g. symptom, therapeutic progress and outcome). The collected data is later compared to data obtained in the same way from patients treated with telemedical support and evaluated regarding differences in the quality of treatment, therapeutic process and the satisfaction of the patients with telemedicine. The aim is to improve the treatment quality in regional hospitals and practices of patients with serious and complex diseases and bring forward the application of telemedicine.

DETAILED DESCRIPTION:
In future time the number of old people will significantly increase in Germany because of the demographic change taking place. The health care of the large number of old people will probably lead to a lack of physicians and an inefficient health care system. One strategy to tackle the problem could be telemedicine. Telemedicine makes it possible to provide know-ledge from experts to local hospitals and practices which otherwise need to send patients with serious and complex diseases to specialized trans-regional health centers. In this multicenter, prospective, non-interventional study hospitals and practices in NRW are supplied via a telematics platform with expert know-ledge from the university hospitals RWTH Aachen and Münster. The communication occurs via highly encrypted audio/video conference systems and a certified data exchange platform "Fallakte+".

In total 40.000 outpatient and stationary patients should be treated with telemedical support. Registered doctors will be involved in already existing practice networks to evaluate the potential for transfer and to ensure the sharing of know-ledge beyond the borders of individual sectors. The aim of the study is to improve the treatment quality of regional hospitals and practices and to increase the efficiency of the care of relevant patient cohort in the field of infectiology and intensive care with the main focus sepsis as those patient groups especially often require professional expertise for a successful therapy.

In the beginning of the study participating hospitals and practices are randomly distributed into four clusters (cluster randomization). The different clusters all start with the control phase but enter into the intervention phase at different times (stepped-wedge design). During the control phase data of patients with infection and intensive care patients routinely treated without the support of telemedicine are documented and the patients are asked to complete a questionnaire regarding health-related quality of life (SF36) directly after treatment and at two time points in the follow-up. The collected data will be later compared to data obtained in the same way from patients treated with telemedical support and evaluated regarding differences in the quality of treatment, therapeutic process and the satisfaction of the patients with telemedicine.

If the study shows that the treatment quality and therapeutic process of patients with infectious diseases or need for intensive care is improved by telemedicine, the telematics platform can be expanded and used by other specialized fields and users in future time.

ELIGIBILITY:
Inclusion Criteria:

* majority
* written informed consent
* infectiological and/or intensive care treatment

Exclusion Criteria:

* minority
* absence of written informed consent in the case of non-acute life-threatening disease
* persons who have a dependency or employment relationship with the sponsor or investigator
* persons who are sheltered in an institution upon court or administrative order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159065 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Improvement of treatment quality | through study completion, an average of 30 days up to a maximum of 1 year
  The level of implementation of the 10 recommendations of the German Society of Infectious Diseases (Deutsche Gesellschaft für Infektiologie, DGI) within the framework of the Initiative "Decide wisely" ("Klug entscheiden").

SECONDARY OUTCOMES:
Rate of sepsis diagnosis | through study completion, an average of 30 days up to a maximum of 1 year
  Rate of sepsis diagnosis
Rate of ARDS Diagnosis | through study completion, an average of 30 days up to a maximum of 1 year
  Rate of ARDS Diagnosis
Sepsis therapy in compliance with guidelines | through study completion, an average of 30 days up to a maximum of 1 year
  Sepsis therapy in compliance with guidelines through for instance timely administration of antibiotics within 3 h and reduction of sepsis mortality.
Rate of ARDS therapy according to guidelines | through study completion, an average of 30 days up to a maximum of 1 year
  Measured against the evident ventilation targets, Ventilation with low ventilation volumes and low peak pressures: with controlled ventilation:
  Breath volume of 6 ml/kg calculated Body ideal weight, PEEP setting in proportion with the necessary FiO2, plateau pressure < 30 cm H2O
Rate of inadequate antibiotic therapies | through study completion, an average of 30 days up to a maximum of 1 year
  Measured by the Percentage of postoperatively continued perioperative Antibiotic prophylaxis
Rate of patients with dialysis | At discharge from Intensive Care Unit (study completion); after an average of 30 days up to a maximum of 1 year
  Rate of patients with dialysis requiring Kidney insufficiency in discharge from the Intensive care
Rate of transfer transport | At discharge from Intensive Care Unit (study completion); after an average of 30 days up to a maximum of 1 year
  Rate of transfer transport
Health-related quality of life (SF36-Questionnaire) | At discharge from Intensive Care Unit (through study completion; an average of 30 days up to a maximum of 1 year), through study completion, an average of 12 months and 24 months after discharge of ICU
  Clinical studies 36-item Medical Outcomes Study Short-Form General Health Survey An instrument used to assess multidimensional health-related QOL, which measures 8 health related parameters: physical function, social function, physical role, emotional role, mental health, energy, pain, general health perceptions; each parameter is scored from 0 to 100 Managed care 36-Item Short-Form Functional and Perceived Health Status Survey A questionnaire which measures health status; the SF-36 also includes a list of 18 self-reported chronic conditions
Rate of non-diagnosed sepsis | through study completion, an average of 30 days up to a maximum of 1 year
  Defined as no filled out sepsis bundle despite presence of sepsis symptoms
Sepsis mortality rate | through study completion, an average of 30 days up to a maximum of 1 year
  Sepsis mortality rate
Hospital mortality rate | through study completion, an average of 30 days up to a maximum of 1 year
  Hospital mortality rate
Length of stay in intensive care unit | At discharge from Intensive Care Unit (study completion); after an average of 30 days up to a maximum of 1 year
  Length of stay in intensive care unit measured in hours
Hospital stay | At discharge from Hospital; after an average of 30 days up to a maximum of 1 year
  Hospital stay measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Gernot Marx, Univ.-Prof. Dr. med., Principal Investigator — Clinic for Operative Intensive Care and Intermediate Care, University Hospital RWTH Aachen
Locations (2):
- Germany (2):
  - University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia
  - University Hospital Münster, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engel C, Brunkhorst FM, Bone HG, Brunkhorst R, Gerlach H, Grond S, Gruendling M, Huhle G, Jaschinski U, John S, Mayer K, Oppert M, Olthoff D, Quintel M, Ragaller M, Rossaint R, Stuber F, Weiler N, Welte T, Bogatsch H, Hartog C, Loeffler M, Reinhart K. Epidemiology of sepsis in Germany: results from a national prospective multicenter study. Intensive Care Med. 2007 Apr;33(4):606-18. doi: 10.1007/s00134-006-0517-7. Epub 2007 Feb 24. PMID 17323051
- [Background] Reinhart K, Brunkhorst FM, Bone HG, Bardutzky J, Dempfle CE, Forst H, Gastmeier P, Gerlach H, Grundling M, John S, Kern W, Kreymann G, Kruger W, Kujath P, Marggraf G, Martin J, Mayer K, Meier-Hellmann A, Oppert M, Putensen C, Quintel M, Ragaller M, Rossaint R, Seifert H, Spies C, Stuber F, Weiler N, Weimann A, Werdan K, Welte T; German Sepsis Society; German Interdisciplinary Association of Intensive Care and Emergency Medicine. Prevention, diagnosis, therapy and follow-up care of sepsis: 1st revision of S-2k guidelines of the German Sepsis Society (Deutsche Sepsis-Gesellschaft e.V. (DSG)) and the German Interdisciplinary Association of Intensive Care and Emergency Medicine (Deutsche Interdisziplinare Vereinigung fur Intensiv- und Notfallmedizin (DIVI)). Ger Med Sci. 2010 Jun 28;8:Doc14. doi: 10.3205/000103. PMID 20628653
- [Background] Laxminarayan R, Bhutta Z, Duse A, Jenkins P, O'Brien T, Okeke IN, Pablo-Mendez A, Klugman KP. Drug Resistance. In: Jamison DT, Breman JG, Measham AR, Alleyne G, Claeson M, Evans DB, Jha P, Mills A, Musgrove P, editors. Disease Control Priorities in Developing Countries. 2nd edition. Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2006. Chapter 55. Available from http://www.ncbi.nlm.nih.gov/books/NBK11774/ PMID 21250349
- [Derived] Marx G, Greiner W, Juhra C, Elkenkamp S, Gensorowsky D, Lemmen S, Englbrecht J, Dohmen S, Gottschalk A, Haverkamp M, Hempen A, Flugel-Bleienheuft C, Bause D, Schulze-Steinen H, Rademacher S, Kistermann J, Hoch S, Beckmann HJ, Lanckohr C, Lowitsch V, Peine A, Juzek-Kuepper F, Benstoem C, Sperling K, Deisz R. An Innovative Telemedical Network to Improve Infectious Disease Management in Critically Ill Patients and Outpatients (TELnet@NRW): Stepped-Wedge Cluster Randomized Controlled Trial. J Med Internet Res. 2022 Mar 2;24(3):e34098. doi: 10.2196/34098. PMID 35103604
- See also: Jung, N. Klug entscheiden: . . . in der Infektiologie. Dtsch Arztebl 2016; 113(13): A-608 / B-514 / C-510 — https://www.aerzteblatt.de/archiv/175621/Klug-entscheiden-in-der-Infektiologie